CLINICAL TRIAL: NCT00050960
Title: Randomized Phase III Trial Comparing Targretin Capsules/Carboplatin/Paclitaxel Versus Carboplatin/Paclitaxel in Chemotherapy-Naïve Patients With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Evaluation of Efficacy, Safety and Tolerability of Targretin Capsules in Patients With Advanced or Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Eisai, Inc, Eisai, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L1069-48; NCT00036907 (obsolete NCT alias)
Record Dates: First submitted 2002-12-31; First posted 2003-01-03 (Estimated); Results first posted 2010-08-24 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Targretin; Retinoid; Bexarotene
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bexarotene; Carboplatin; Paclitaxel

ARMS (2):
- bexarotene with carboplatin and paclitaxel (Experimental)
  Interventions: Drug: bexarotene with carboplatin and paclitaxel
- carboplatin and paclitaxel (Experimental)
  Interventions: Drug: carboplatin and paclitaxel

INTERVENTIONS:
Drug: bexarotene with carboplatin and paclitaxel — bexarotene capsules (400 mg/m^2/day) in combination with carboplatin IV (AUC 6) every 3 weeks and paclitaxel IV (200 mg/m^2) every 3 weeks. Subjects in this group also received an antilipid agent which was selected at the discretion of the investigator.
  Arms: bexarotene with carboplatin and paclitaxel
Drug: carboplatin and paclitaxel — carboplatin IV (AUC 6) every 3 weeks and paclitaxel IV (200 mg/m^2) every 3 weeks.
  Arms: carboplatin and paclitaxel

SUMMARY:
This study evaluates the use of Targretin capsules (bexarotene) in combination with standard chemotherapy for the treatment of metastatic Non-Small Cell Lung Cancer (NSCLC) in patients who have not yet received chemotherapy for their lung cancer.

DETAILED DESCRIPTION:
This study evaluates the use of Targretin capsules (bexarotene) in combination with Carboplatin and Paclitaxel for the treatment of metastatic non-small cell lung cancer in patients who have not yet received chemotherapy for their lung cancer. Every patient receives a platinum-containing chemotherapy every three weeks for at least four chemotherapy cycles (approximately four months). Half of the patients are randomly assigned to receive Targretin capsules once daily in addition to the chemotherapy. The other half is randomized to receive a standard platinum-containing chemotherapy without Targretin capsules.

ELIGIBILITY:
Patients must have:

* Pathologic (histologic or cytologic) confirmation of NSCLC
* Stage IIIB with malignant pleural effusion or Stage IV disease
* At least one measurable or evaluable NSCLC lesion that has not been previously irradiated unless radiation therapy was more than three weeks prior to entry in the study and the lesion has been shown to have progressed subsequent to the radiation therapy
* ECOG performance status 0 or 1
* Adequate organ system function
* Fasting serum triglycerides that are within the age-adjusted normal range (or normalized with appropriate intervention such as antilipid therapy prior to the initiation of Targretin capsule therapy).

Patients must be able to complete at least four cycles of combination chemotherapy (i.e., approximately four months)

Patients must not have had:

* Brain metastasis
* Prior chemotherapy for NSCLC
* Prior platinum-based chemotherapy for any indication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2002-05; Primary Completion 2004-07 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mack Mabry, M.D., Study Director — Ligand Pharmaceuticals
Locations (154):
- United States (121):
  - Montgomery Cancer Center, L.L.C., Montgomery, Alabama
  - Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Bay Area Cancer Research Group, LLC, Concord, California
  - Compassionate Cancer Care Medical Group, Inc., Fountain Valley, California
  - Pacific Coast Hematology/Oncology Medical Group, Inc., Fountain Valley, California
  - California Cancer Care, Inc., Greenbrae, California
  - Coast Hematology and Oncology Associates, Long Beach, California
  - Metropolitan Hematology/Oncology Medical Group, Los Angeles, California
  - Sant P. Chawla, Inc., Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Sutter Gould Medical Foundation, Modesto, California
  - Medical Oncology Care Associates, Orange, California
  - Southern California Kaiser Permanente Medical Group, San Diego, California
  - Sharp Health Care, San Diego, California
  - UCSF/Mount Zion Comprehensive Cancer Center, San Francisco, California
  - Medical Group of North County, Inc., San Diego Cancer Center, Vista, California
  - Rocky Mountain Cancer Centers - Midtown, Denver, Colorado
  - Eastern Connecticut Hematology & Oncology, Norwich, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Comprehensive Cancer Care Specialists of Boca Raton, Boca Raton, Florida
  - University of Florida/Jacksonville, Jacksonville, Florida
  - Watson Clinic, Lakeland, Florida
  - Oncology and Radiation Associates, Miami, Florida
  - Florida Cancer Institute, New Port Richey, Florida
  - Florida Oncology Associates, Orange Park, Florida
  - Cancer Centers of Florida, P.A., Orlando, Florida
  - South Florida Oncology & Hematology Consultants, Plantation, Florida
  - Medical Oncology Associates of Augusta, Augusta, Georgia
  - Georgia Oncology Partners Research & Education Foundation, Marietta, Georgia
  - St. Luke's/Mountain State Tumor Institute (MSTI), Boise, Idaho
  - Weiss Memorial Hospital, Chicago, Illinois
  - Northwest Oncology and Hematology, SC, Elk Grove Village, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Hematology Oncology Assoc. of Illinois, Skokie, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Cancer Care Center, New Albany, Indiana
  - Michiana Hematology-Oncology, South Bend, Indiana
  - Kansas City Oncology and Hematology Group, Kansas City Cancer Centers, Overland Park, Kansas
  - Drs. Carroll, Sheth, and Raghavan, Louisville, Kentucky
  - Southwest Oncology Associates, Lafayette, Louisiana
  - APMC, Metairie, Louisiana
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Chesapeake Oncology-Hematology Associates, Baltimore, Maryland
  - Associates in Oncology/Hematology PC, Rockville, Maryland
  - Berkshire Hematology Oncology, PC, Pittsfield, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Providence Cancer Institute, Southfield, Michigan
  - St. Lukes Hospital, Duluth, Minnesota
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Hematology Oncology Centers of the Northern Rockies, Billings, Montana
  - Montana Cancer & Infectious Disease Specialists, Missoula, Montana
  - Cancer and Blood Specialists of Nevada, Henderson, Nevada
  - Nevada Cancer Center, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Orange Medical Group, East Orange, New Jersey
  - VA New Jersey Health Care System, East Orange, New Jersey
  - Hematology-Oncology Associates of Northern NJ, PA, Morristown, New Jersey
  - Somerset Hematology Oncology Associates, Somerset, New Jersey
  - University of Medicine & Dentistry of NJ, School of Osteopathic Medicine, Stratford, New Jersey
  - Overlook Oncology Center, Summit, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - New York Oncology Hematology, P.C., Capital District Hematology Oncology Associates, Albany, New York
  - Erie Medical Center, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Arena Oncology Associates, Great Neck, New York
  - Cancer Institute of Long Island, Inc., Great Neck, New York
  - Cancer Research of Long Island, Inc., Great Neck, New York
  - Broome Oncology, LLC, Johnson City, New York
  - New York Presbyterian Hospital, Weill Medical College of Cornell University, New York, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - VA Medical Center, Northport, New York
  - New York Oncology Hematology, P.C., Riverview Cancer Care Medical Associates, Rexford, New York
  - South Shore Hematology Oncology Associates, PC, Rockville Centre, New York
  - Raleigh Hematology Oncology Clinic, Cary, North Carolina
  - Northwest Carolina Oncology and Hematology, P.A., Hickory, North Carolina
  - Nashat Y. Gabrail, MD, Inc., Canton, Ohio
  - University of Cincinnati, Barrett Cancer Center, Cincinnati, Ohio
  - Columbus Community Clinical Oncology Program, Columbus, Ohio
  - Dayton Oncology/Hematology Consultants, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Oncology/Hematology, Kaiser Permanente Northwest, Portland, Oregon
  - Oncology Hematology of Lehigh Valley, PC, Bethlehem, Pennsylvania
  - Medical Oncology Associates of Wyoming Valley, PC, Kingston, Pennsylvania
  - Charleston Hematology Oncology P.A., Charleston, South Carolina
  - Liberty Hematology/Oncology, Columbia, South Carolina
  - WJB Dorn VA Medical Center, Columbia, South Carolina
  - Cancer Centers of the Carolinas, Seneca, South Carolina
  - Santee Hematology/Oncology, Sumter, South Carolina
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Boston Baskin Cancer Group, Memphis, Tennessee
  - Texas Oncology, P.A., Arlington, Texas
  - South Austin Cancer Center, Austin, Texas
  - Lone Star Oncology Consultants, P.A., Austin, Texas
  - Cancer Specialists of South Texas, PA, Corpus Christi, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - Texas Oncology, P.A., Garland, Texas
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Allison Cancer Center, Midland, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Hope Oncology, Richardson, Texas
  - Hematology & Oncology Associates of South Texas, San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texoma Cancer Center, Wichita Falls, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Arlington Fairfax Hematology Oncology, Arlington, Virginia
  - Hematology Oncology Patient Enterprises, Center for Cancer Care, Charlottesville, Virginia
  - Danville Hematology & Oncology, Inc., Danville, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Stark MD, PC, Portsmouth, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Yakima Regional Cancer Care Center, Internal Medicine Associates of Yakima, Inc., Yakima, Washington
  - Morgantown Internal Medicine Group, Morgantown, West Virginia
- Austria (3):
  - Sozialmedizinisches Zentrum, Vienna
  - Kaiser-Franz-Josef-Spital, Vienna
  - Allgemeines offentliches Krankenhaus der barmherzigen Schwestern vom Heiligen Kreuz Pneumologie, Wels
- Canada (3):
  - Algoma Regional Cancer Program - Sault Area Hospital, Sault Ste. Marie, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - S.M.B.D. Jewish General Hospital, Montreal, Quebec
- France (15):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Centre Hospitalier General de la Region Annecienne, Annecy
  - Centre Hospitalier d'Antibes-Juan-Les-Pins, Antibes
  - CHRU Hopital de Bois Guillaume, Bois-Guillaume
  - DOP International, Créteil
  - Hopital de Draguignan, Draguignan
  - Centre Hospitalier General, Gap
  - Hopital du Cluzeau, Limoges
  - CHU Hopital St. Marguerite, Marseille
  - Centre Regional de Lutte contre le Cancer (CRLC), Val d'Aurelle-Paul Lamarque, Montpellier
  - Hopital Saint Antoine, Paris
  - CHU - Hopital Nord, Saint-Etienne
  - Hopital Saint Anne, Toulon Naval
  - Service de Pneumology, Hopital Adulte de Brabois, Vandœuvre-lès-Nancy
  - Centre Hospitalier, Villefranche Sur Soane
- Germany (5):
  - Dept. of Internal Medicine, St. Nikolaus-Stiftshospital Andernach, Andernach
  - Aesklepios-Fachkliniken Muchen-Gauting, Gauting
  - Krankenhaus GroBhansdorf, Zentrum fur Pneumologie und Thoraxchirurgie, GroBhansdorf
  - Ludwig-Maximilians Universitat Munchen, München
  - Charite Universitatsklinikum der Humboldt-Universitat zu Berlin, SchumannstraBe, Berlin
- Spain (7):
  - Hospital Provincial de Castellon, Castellon
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitario La Fe Servicio de Oncologia, Valencia
  - Hospital Arnau de Villanova, Servicio de Oncologia, Valencia
  - Hospital Clinico Universitario, Servicio Hematologia y Oncologia, Valencia
  - Hospital de Sagunto Servicio de Oncologia, Valencia

REFERENCES:
- See also: Related Info — http://www.Ligand.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bexarotene With Carboplatin and Paclitaxel | Carboplatin and Paclitaxel
Started | 306 | 306
Completed | 4 (Represents number of patients with no primary reason for termination) | 2 (Represents number of patients with no primary reason for termination)
Not Completed | 302 | 304
Not completed — Progressive Disease | 137 | 93
Not completed — Stable Disease | 19 | 48
Not completed — Partial Response | 14 | 19
Not completed — Complete Response | 0 | 2
Not completed — Adverse Event | 62 | 61
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 23 | 18
Not completed — Administrative | 31 | 46
Not completed — Non-compliance | 3 | 1
Not completed — Death | 13 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bexarotene With Carboplatin and Paclitaxel | Carboplatin and Paclitaxel | Total
Number analyzed (Participants) | 306 | 306 | 612
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 166 | 174 | 340
  >=65 years | 140 | 132 | 272
Age Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.6) | 61.7 (10.3) | 62.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 103 | 206
  Male | 203 | 203 | 406
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 9 | 11
  Not Hispanic or Latino | 304 | 297 | 601
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Number; unit: Participants] — Counts are correct as reported. The BL measure title of "race" does not include counts of Hispanic or Latino population- which are reported in the BL measure title of "Ethnicity."
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 7 | 3 | 10
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 23 | 20 | 43
    White | 269 | 272 | 541
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: From date of randomization to date of death
Population: Intent-to-Treat (ITT)
Measure: Median (Full Range); unit: Months
Arm/Group | Bexarotene With Carboplatin and Paclitaxel | Carboplatin and Paclitaxel
Number analyzed (Participants) | 306 | 306
Months | 8.5 [7.7 to 9.3] | 9.2 [8.3 to 10.5]

ADVERSE EVENTS:
Description: Number of participants at risk reflects the number exposed to at least one dose of any study medication. Twenty-four subjects in Participant Flow did not receive any study medication.
Arm/Group | Bexarotene With Carboplatin and Paclitaxel | Carboplatin and Paclitaxel
Serious Adverse Events (participants affected / at risk) | 256/293 | 242/295
Other Adverse Events (participants affected / at risk) | 293/293 | 295/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bexarotene With Carboplatin and Paclitaxel (N=293) | Carboplatin and Paclitaxel (N=295)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 219 | 213
Non-small cell lung cancer Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 19 | 7
Anorexia (Metabolism and nutrition disorders) | 4 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 11
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Anaemia (Blood and lymphatic system disorders) | 14 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 11 | 9
Neutropenia (Blood and lymphatic system disorders) | 11 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 4
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 9 | 6
Nausea (Gastrointestinal disorders) | 8 | 6
Diarrhea (Gastrointestinal disorders) | 8 | 5
Abdominal pain (Gastrointestinal disorders) | 5 | 1
Constipation (Gastrointestinal disorders) | 4 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 4
Cardiac failure congestive (Cardiac disorders) | 1 | 4
Pericardial effusion (Cardiac disorders) | 1 | 3
Pyrexia (General disorders) | 12 | 8
Asthenia (General disorders) | 9 | 4
Chest pain (General disorders) | 3 | 7
Fatigue (General disorders) | 3 | 1
Oedema peripheral (General disorders) | 3 | 1
Pain (General disorders) | 3 | 1
Hepatic failure (Hepatobiliary disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Pneumonia (Infections and infestations) | 9 | 6
Sepsis (Infections and infestations) | 3 | 2
Convulsion (Nervous system disorders) | 4 | 3
Cerebrovascular accident (Nervous system disorders) | 3 | 1
Spinal cord compression (Nervous system disorders) | 4 | 0
Polyneuropathy (Nervous system disorders) | 3 | 1
Confusional state (Psychiatric disorders) | 4 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 7
Hypotension (Vascular disorders) | 2 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bexarotene With Carboplatin and Paclitaxel (N=293) | Carboplatin and Paclitaxel (N=295)
Anemia (Blood and lymphatic system disorders) | 147 | 112
Neutropenia (Blood and lymphatic system disorders) | 138 | 71
Thrombocytopenia (Blood and lymphatic system disorders) | 44 | 42
Leukopenia (Blood and lymphatic system disorders) | 31 | 12
Febrile neutropenia (Blood and lymphatic system disorders) | 17 | 10
Hypotriglyceridemia (Metabolism and nutrition disorders) | 168 | 6
Anorexia (Metabolism and nutrition disorders) | 71 | 48
Dehydration (Metabolism and nutrition disorders) | 40 | 22
Hypercholesterolemia (Metabolism and nutrition disorders) | 35 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 26 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 22 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 8
Hyponatremia (Metabolism and nutrition disorders) | 16 | 6
Hyperlipidemia (Metabolism and nutrition disorders) | 16 | 2
Insomnia (Psychiatric disorders) | 70 | 56
Depression (Psychiatric disorders) | 39 | 27
Anxiety (Psychiatric disorders) | 32 | 31
Confusional state (Psychiatric disorders) | 24 | 7
Neuropathy peripheral (Nervous system disorders) | 69 | 70
Dizziness (Nervous system disorders) | 44 | 32
Headache (Nervous system disorders) | 38 | 28
Paraesthesia (Nervous system disorders) | 29 | 34
Polyneuropathy (Nervous system disorders) | 28 | 31
Neuropathy (Nervous system disorders) | 26 | 19
Dysgeusia (Nervous system disorders) | 17 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 74 | 52
Cough (Respiratory, thoracic and mediastinal disorders) | 61 | 47
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 20 | 23
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 17 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 | 11
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 9
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 15 | 10
Hypotension (Vascular disorders) | 18 | 10
Flushing (Vascular disorders) | 16 | 9
Nausea (Gastrointestinal disorders) | 147 | 140
Diarrhoea (Gastrointestinal disorders) | 108 | 68
Vomiting (Gastrointestinal disorders) | 96 | 78
Constipation (Gastrointestinal disorders) | 80 | 84
Abdominal pain (Gastrointestinal disorders) | 39 | 19
Dyspepsia (Gastrointestinal disorders) | 19 | 19
Stomatitis (Gastrointestinal disorders) | 19 | 18
Abdominal pain upper (Gastrointestinal disorders) | 17 | 12
Dysphagia (Gastrointestinal disorders) | 20 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 147 | 154
Rash (Skin and subcutaneous tissue disorders) | 47 | 22
Pruritis (Skin and subcutaneous tissue disorders) | 27 | 20
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 35 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 24 | 5
Skin desquamation (Skin and subcutaneous tissue disorders) | 15 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 78 | 68
Myalgia (Musculoskeletal and connective tissue disorders) | 61 | 55
Pain in extremity (Musculoskeletal and connective tissue disorders) | 55 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 34 | 35
Bone pain (Musculoskeletal and connective tissue disorders) | 23 | 16
Fatigue (General disorders) | 156 | 137
Asthenia (General disorders) | 67 | 49
Chest pain (General disorders) | 44 | 56
Oedema peripheral (General disorders) | 39 | 38
Pain (General disorders) | 27 | 30
Pyrexia (General disorders) | 46 | 47
Weight decreased (Investigations) | 41 | 30
Blood triglycerides increased (Investigations) | 27 | 0
Hypothyroidism (Endocrine disorders) | 73 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No